CLINICAL TRIAL: NCT05053698
Title: Evolution of Aqueous Flare in Rhegmatogenous Retinal Detachments Treated With Gas or Silicone Oil Tamponade.
Acronym: FLADESIL
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BERROD Jean-Paul, Professor BERROD Jean-Paul, Central Hospital, Nancy, France
Other Study IDs: 2020PI209
Record Dates: First submitted 2021-06-04; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Retinal Detachment
Keywords: Aqueous Flare; Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Initial gas tamponade: Primary vitrectomy and fluid-air exchange with SF6 or C2F6 gas tamponade
  Interventions: Other: Aqueous flare measurement
- Initial silicone oil tamponade: Primary vitrectomy and fluid-air exchange with silicone oil tamponade
  Interventions: Other: Aqueous flare measurement
- Relapse treated with gas tamponade: Secondary vitrectomy and fluid-air exchange with SF6 or C2F6 or C3F8 gas tamponade
  Interventions: Other: Aqueous flare measurement
- Relapse treated with silicone oil tamponade: Secondary vitrectomy and fluid-air exchange with silicone oil tamponade
  Interventions: Other: Aqueous flare measurement

INTERVENTIONS:
Other: Aqueous flare measurement — Aqueous flare was measured preoperatively and postoperatively with a laser flare-cell meter (LFCM ; Kowa FM-500, Kowa Company Ltd, Tokyo, Japan).

SUMMARY:
To examine and to compare the evolution of aqueous flare from presentation until the third postoperative month in a series of consecutive patients who underwent primary vitrectomy for rhegmatogenous retinal detachment (RRD), in 4 groups of patients :

* Group 1 : 48 eyes primarily treated with gas tamponade
* Group 2 : 11 eyes primarily treated with silicone oil tamponade
* Sub-Group G1RG : 8 eyes among Group 1 treated with gas after relapse
* Sub-Group G1RS : 3 eyes among Group 1 treated with silicone oil after relapse

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* patients who underwent surgery for rhegmatogenous retinal detachment (silicone or gas tamponade)
* aqueous flare measurement carried out preoperatively and postoperatively at 2-4 weeks and 3 months

Exclusion Criteria:

* diabetic retinopathy
* glaucoma
* non rhegmatogenous retinal detachment
* active uveitis
* pseudoexfoliation syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients addressed at the Ophthalmology Department for Rhegmatogenous Retinal Detachment and who matched the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Change in aqueous flare measurement (expressed as photon counts per millisecond and measured with a laser flare-cell meter) | preoperatively and postoperatively at 2 weeks and 3 months after surgery
  Aqueous flare was measured preoperatively and postoperatively at 2 weeks, 4 weeks and 3 months with a laser flare-cell meter, in patients treated for RRD

SECONDARY OUTCOMES:
Change in aqueous flare measurement (measured with a laser flare-cell meter) | postoperatively at 2 weeks and 3 months after surgery
  To describe the evolution of the aqueous humor flare between the postoperative visits at 2 weeks and at 3 months after retinal detachment surgery in each groups of patients.
Comparison of aqueous flare values (measured with a laser flare-cell meter) between patients who relapsed and patients who didn't relapse | preoperative
  To compare the preoperative flare measurements between patients without versus with recurrence among those treated with gas
Evolution of measures of visual acuity | preoperatively and postoperatively at 3 months
  The best-corrected visual acuity (BCVA) was measured with projected-light Snellen charts and expressed in logMAR.
Evolution of macular status | preoperatively and postoperatively at 3 months
  Evaluation of macular status with macular imaging by optical coherence tomography (Heidelberg Engineering)
Relapsing status (yes or not) | at 3 months postoperative
  Determined by careful fundus and peripheral retina examination.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul BERROD, Professor MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- BERROD Jean-Paul MD, Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No